CLINICAL TRIAL: NCT06713551
Title: The Effect of Big Amplitude Calisthenic Group Exercises With Music on Balance and Dual Task Performance in Elderly Individuals
Brief Title: The Effect of Big Amplitude Calisthenic Group Exercises on Balance and Dual Task Performance in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Guzin Kaya Aytutuldu, Assistant Professor, Biruni University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BiruniU.
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Older People
Keywords: exercise; high amplitude; music therapy; older adults
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Big amplitude calisthenic group exercises with music (Experimental): The exercise program will consist of balance and mobility-oriented exercises such as reaching forward and upward while sitting on a chair, taking steps forward, backward, sideways and backward while standing, transferring weight, counting in place, sit-to-stand exercises, walking, changing directions or walking over obstacles (Appendix: Exercise Program). This exercise program will be applied to the first group with the accompaniment of classical Western music, while the other group will be applied without music. The exercise programs will be performed for both groups for 40 minutes, two days a week and for eight weeks.
  Interventions: Other: Big Amplitude Calisthenic Group Exercise with Music
- Big amplitude calisthenic group exercises (Active Comparator): The exercise program will consist of balance and mobility-oriented exercises such as reaching forward and upward while sitting on a chair, taking steps forward, backward, sideways and backward while standing, transferring weight, counting in place, sit-to-stand exercises, walking, changing directions or walking over obstacles (Appendix: Exercise Program). This exercise program will be applied to the first group with the accompaniment of classical Western music, while the other group will be applied without music. The exercise programs will be performed for both groups for 40 minutes, two days a week and for eight weeks.
  Interventions: Other: Big Amplitude Calisthenic Group Exercise

INTERVENTIONS:
Other: Big Amplitude Calisthenic Group Exercise with Music — The exercise program will consist of balance and mobility-oriented exercises such as reaching forward and upward while sitting on a chair, taking steps forward, backward, sideways and backward while standing, transferring weight, counting in place, sit-to-stand exercises, walking, changing directions or walking over obstacles (Appendix: Exercise Program). This exercise program will be applied to the first group with the accompaniment of classical Western music, while the other group will be applied without music. The exercise programs will be performed for both groups for 40 minutes, two days a week and for eight weeks.
  Arms: Big amplitude calisthenic group exercises with music
Other: Big Amplitude Calisthenic Group Exercise — The exercise program will consist of balance and mobility-oriented exercises such as reaching forward and upward while sitting on a chair, taking steps forward, backward, sideways and backward while standing, transferring weight, counting in place, sit-to-stand exercises, walking, changing directions or walking over obstacles (Appendix: Exercise Program). This exercise program will be applied to the first group with the accompaniment of classical Western music, while the other group will be applied without music. The exercise programs will be performed for both groups for 40 minutes, two days a week and for eight weeks.
  Arms: Big amplitude calisthenic group exercises

SUMMARY:
The subject of this research is to investigate the effect of high amplitude calisthenic group exercises with music on balance and dual task performance in elderly individuals.

The aim of this study is to examine the effect of music during high amplitude calisthenic group exercises on dual task performance and balance in elderly residents living under the administration of Kagıthane Municipality in Istanbul.

DETAILED DESCRIPTION:
Old age represents the final stage of human life, an inevitable process of aging that leads to functional and physical impairments. The World Health Organization (WHO) defines old age as "a decrease in the capacity to adapt to environmental factors." Aging is characterized by a decline in fertility, increased mortality, and disability, alongside progressive loss of function. Balance problems are common among the elderly. During motor activities, there is a limited support area that can cause changes in the body's center of gravity. As long as the center of gravity remains within this area, movement can be maintained without disruption. Reduced sensory input and sensitivity in the elderly affect movement clarity and postural stability. This condition necessitates the development of movement strategies that limit the support area to a narrower space and require more accurate control of the center of gravity position. As the center of gravity shifts toward the limits, the likelihood of balance loss increases. Therefore, in order to maintain a safe balance area, circular and forward-backward swing amplitudes decrease in the elderly. During these swings, the elderly must keep the center of pressure on the feet close to stability limits. It is reported that physically active elderly individuals exhibit less anxiety and stress compared to sedentary individuals, and have higher quality of life.Physiotherapy methods focus on improving reaction speed to unexpected perturbations through ankle, hip, and stepping strategies in balance training. Dual task exercises are one of the physiotherapy methods used in balance training. Dual Task In daily life, we rarely perform only one task at a time. Rather, our daily activities often involve performing two or more tasks simultaneously. This is referred to as dual-tasking, for example, searching for something in a pocket while walking, or walking while talking involves dual-task performance. Dual-tasking is based on dividing attention between two simultaneous tasks. Given that attention is a limited resource, dividing attention between two concurrent tasks can lead to a decrease in performance in either or both tasks, especially when the demands of one task are high. The relative change in performance associated with dual tasking is called dual task interference or dual task effect. There are some paradigms that explain dual tasking. The complex nature of processes related to dual tasking is evaluated using these paradigms; here, there are two tasks that are simultaneously performed without any manipulation of task variables, and no instruction is given regarding task priority. It is generally used to investigate dual tasking in each of the two simultaneous tasks. In older individuals, there is a decrease in walking speed during dual tasking due to impairment in executive functions and working memory. The decrease in walking speed during dual tasking in older adults has been shown to be more often associated with cognitive function impairment compared to young adults. In a case study, it was shown that balance exercises performed with dual tasking yielded better results in balance parameters compared to balance exercises performed with single tasking, and longer-lasting results were achieved. Music therapy, defined as "the clinical and evidence-based use of music interventions in a therapeutic relationship to achieve personalized goals completed by a certified professional who has completed an approved music therapy program," can be an effective non-pharmacological treatment method. De Witte and colleagues' meta-analysis found that music interventions had a significant impact on reducing both physiological and psychological stress in 104 RCT music intervention studies involving 9617 participants. To our knowledge, there is no study investigating the effect of high amplitude calisthenic group exercises with music on balance and dual task performance in elderly individuals. Therefore, the study will investigate the effectiveness of an exercise program with music applied in groups, comparing the results between groups.

Scientific studies conducted on the elderly indicate that dual task training has benefits in improving walking, balance, and mobility performance in healthy elderly individuals. In rehabilitation, dual task training has been concluded to be included in preventive physiotherapy approaches for preventing falls and supporting a more active lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* To receive at least 21 points from the Mini Mental Test Evaluation
* To reside in the region affiliated with the Kağıthane Municipality
* To be independent in daily living activities
* To have access to the Kağıthane Municipality Elderly Day Service Center

Exclusion Criteria:

* Having vision and hearing problems
* Neurological, orthopedic problems
* Accompanying cardiovascular problems
* Using a walking aid

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-11-27 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Mini-Best Test | 10 minutes
  The main focus of the Mini-BEST TEST is to emphasize dynamic balance. The scale is used to assess balance and the risk of falling. It allows for the dynamic assessment of balance. It consists of 14 task items representing four balance control systems: prospective posture adjustments, compensatory postural adjustments, sensory orientation, and walking stability. Some tasks involve sitting; these are standing, standing on tiptoe, single-leg standing, compensatory reactions forward, backward, and sideways, tasks to be performed with eyes closed on a sloping surface with foam surface and walking. Speed changes, dizziness, walking over obstacles, and timing are included. Each item is scored on a three-point scale (0-2), with a total maximum score of 28 points. Better balance performance is indicated by higher scores. 2 points indicate the highest functional level, while 0 indicates the lowest functional level. If a person needs physical assistance to perform, one function gets 0 points.
Dual Task Questionnaire | 7 minutes
  Dual task (DT) is a simultaneous neurophysiological experimental procedure that requires an individual to perform two tasks. DT is also mutual communication between motor and cognitive. When two tasks are performed simultaneously, attention capacity should be used effectively, and attention should be divided according to difficulty and priority. Problems will arise when the difficulty level increases or attention capacity decreases. Evaluation of individuals' DT performance is carried out by clinical tests and laboratory measurements. During these tests, additional tasks such as motor (pressing a button, moving something...) or cognitive (counting, answering simple questions...) tasks are given to the person. Changes in strategies during DT are also examined with varying visual and sensory perception. It will be used to learn dual task performance in the study
Timed Up and Go Test | 5 minutes
  The Timed Up and Go Test is performed by giving verbal instructions to the patient to get up from the chair as quickly and safely as possible, walk 3 meters following the marked line on the floor, turn, walk back again, and sit down. Below 10 seconds; the patient walks independently, the risk of falling is very low. 11-19 seconds; the patient walks independently, there is a low to moderate risk of falling. 20-29 seconds; occasional assistance may be needed, there is a moderate to high risk of falling. Over 30 seconds occasionally, assistance is needed and the risk of falling is high
Geriatric Depression Scale | 7 minutes
  The Geriatric Depression Scale consists of 30 self-reported questions that elderly individuals can easily mark with yes or no responses. Questions 3, 4, 5, 6, 8, 10, 11, 12, 13, 14, 16, 17, 18, 20, 22, 23, 24, 25, 26, and 28 contain reverse statements. In scoring the scale, 1 point is given for each response indicating depression, and 0 points for other responses, which is considered as the total depression score. The scoring of the scale is as follows: 0-10 points "no depression", 11-13 points "possible depression", 14 and above points "definite depression". The scale scores range from a minimum of 1 to a maximum of 30. The evaluation of the Geriatric Depression Scale is as follows: for questions 1, 2, 7, 9, 15, 19, 21, 27, 29, and 30, 1 point is given for each "no" response and 0 points for "yes" response, for questions 3, 4, 5, 6, 8, 10, 11, 12, 13, 14, 16, 17, 18, 20, 22, 23, 24, 25, 26, and 28, 1 point is given for each "yes" response and 0 points for "no" response

SECONDARY OUTCOMES:
Physical Activity Scale for the Elderly (PASE) | 10 minutes
  The Physical Activity Scale for the Elderly (PASE) is a short and applicable scale widely used in the literature, shown to be valid and reliable. The survey assesses the physical activities of elderly individuals in the previous week, covering the physical components of leisure, home, and occupational activities. Leisure activities, light, moderate, and strenuous sports, recreational activities, and muscle strength exercises include the frequency of outdoor walking activities is rarely (1-2 days a week), sometimes (3-4 days a week) and frequent (5 to 7 days a week), and the duration of activities is classified as less than 1 hour, 1 hour to 2 hours, 2 hours to 4 hours, and more than 4 hours.
Mini Mental State Examination | 10 minutes
  Mini Mental State Examination was developed in 1975 to quantitatively assess cognitive impairment in adults. It is a short, convenient, and standardized assessment method that can be used to detect cognitive levels. It consists of a total of 11 items under five main headings: orientation, registration memory, attention and calculation, recall, and language, and is evaluated on a total of 30 points. In the evaluation, 24-30 points indicate normal cognitive function, 18-23 points indicate mild cognitive impairment; 18 points and below indicate a significant impairment of cognitive status.

CONTACTS AND LOCATIONS:
Overall Officials: Guzin Kaya Aytutuldu, Principal Investigator — Biruni University
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colcombe S, Kramer AF. Fitness effects on the cognitive function of older adults: a meta-analytic study. Psychol Sci. 2003 Mar;14(2):125-30. doi: 10.1111/1467-9280.t01-1-01430. PMID 12661673
- [Background] Silsupadol P, Siu KC, Shumway-Cook A, Woollacott MH. Training of balance under single- and dual-task conditions in older adults with balance impairment. Phys Ther. 2006 Feb;86(2):269-81. PMID 16445340
- [Background] de Witte M, Spruit A, van Hooren S, Moonen X, Stams GJ. Effects of music interventions on stress-related outcomes: a systematic review and two meta-analyses. Health Psychol Rev. 2020 Jun;14(2):294-324. doi: 10.1080/17437199.2019.1627897. Epub 2019 Jul 15. PMID 31167611